CLINICAL TRIAL: NCT07163533
Title: Combined Effect of Kendall Exercises With Wearable Vibrotactile Feedback Sensor in Forward Head Posture
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: anees arshad
Record Dates: First submitted 2025-09-01; First posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Neck Pain
Keywords: Forward head posture (FHP); Vibrotactile feedback sensors; Kendall exercises; Craniovertebral angle; Inertial measure units
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Single (Outcomes Assessor) no
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A ( wearable sensors plus kendall exercises ) (Experimental): this group will receives wearable sensors plus Kendall exercises for 4 weeks
  Interventions: Other: wearble vibrotactile feedback sensor and kendel exercises
- group B (kendall exercises only ) (Active Comparator): this group will receives Kendall exercises for 4 weeks
  Interventions: Other: kendel exercises

INTERVENTIONS:
Other: wearble vibrotactile feedback sensor and kendel exercises — Wearable vibrotactile feedback sensor will be applied to the neck for assessment and management and secondly kendel exercises consisting of Strengthening of Deep Cervical Flexors, Stretching the Cervical Extensors, Strengthening Shoulder Retraction, Stretching the Pectoralis Muscle. each exercise will be given 3 days per week for 30 min each.
  Arms: group A ( wearable sensors plus kendall exercises )
Other: kendel exercises — kendel exercises consisting of Strengthening of Deep Cervical Flexors, Stretching the Cervical Extensors, Strengthening Shoulder Retraction, Stretching the Pectoralis Muscle. each exercise will be given 3 days per week for 30 min each.
  Arms: group B (kendall exercises only )

SUMMARY:
The aim of this research is to determines Combined Effect of Kendall exercises with Wearable vibrotactile feedback Sensor on Forward Head Posture correction on neck pain, and improving craniovertebral angle and muscle thickness. Randomized controlled trials at Fauji Foundation Hospital and Margalla Institute of health sciences . The sample size was 64. The subjects were divided in two groups, 32 subjects will be included in wearbable sensors and kendall exercises group and 32 will be in Kendell exercise alone . Study duration will be 12 months. Sampling technique applied will be non probability convinience sampling technique. Participants eligible for recruitment in this study will include young adults between the ages of 18 and 30 years. Eligible participants must also present with a craniovertebral angle (CVA) of less than 50 degrees, a body mass index (BMI) within the range of 18.5-30 kg/m², and a daily screen time of less than five hours. Data will be analyzed through SPSS version 26.

DETAILED DESCRIPTION:
Forward Head Posture (FHP) is one of the most prevalent postural deviations among young adults, largely influenced by prolonged screen use, sedentary behaviors, and faulty sitting postures. This malalignment, characterized by anterior displacement of the head relative to the shoulder line, places excessive strain on the cervical spine and is strongly associated with neck pain, reduced craniovertebral angle (CVA), and muscular imbalances. If not corrected, FHP may contribute to long-term musculoskeletal dysfunction and impaired quality of life.

Conventional corrective approaches, such as the Kendall Exercise protocol, are widely recognized for addressing FHP by stretching shortened muscles (cervical extensors, pectorals) and strengthening weakened stabilizers (deep cervical flexors, scapular retractors). However, exercise-based interventions alone often face challenges of adherence and lack of postural awareness during daily activities.

Wearable vibrotactile feedback sensors have emerged as an innovative adjunct to exercise therapy. These devices provide real-time postural biofeedback, alerting users immediately when deviations occur and actively engaging them in maintaining correct alignment. By combining the Kendall Exercise protocol with wearable biofeedback technology, a more comprehensive approach may be achieved, addressing both neuromuscular strengthening and behavioral postural awareness.

Despite the increasing prevalence of FHP in young adults, limited evidence exists on the combined effect of structured exercise and wearable sensors. No randomized controlled trial has yet evaluated this integrated approach in this population. To address this gap, the present study will assess the combined effect of Kendall exercises and a wearable vibrotactile feedback sensor on forward head posture, neck pain, craniovertebral angle, and cervical muscle thickness in young adults.

ELIGIBILITY:
Inclusion Criteria:

Young Adult with age Between 18 to 30 years Both gender craniovertebral angle (CVA) < 50 degrees BMI 18.5-30 kg/m2 Screen time less than 5 hours/day

Exclusion Criteria:

History of recent neck or spinal surgery (within the past 6 12 months). Diagnosed musculoskeletal, neurological, or vestibular disorders affecting posture, balance, or neck movement (e.g., cervical radiculopathy, scoliosis, Parkinson's, etc.).

Diagnosed Temporomandibular dysfunction Use of assistive devices (e.g., neck brace, posture correctors) in the past 3 months.

Any cognitive or psychological condition that may affect compliance with instructions or accurate reporting of symptoms.

Ongoing participation in a structured exercise or physiotherapy program targeting posture or neck muscles.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
neck pain | baseline to fourth week
  NPRS(0 to 10) 0 means no pain and 10 means severe pain
muscle thickness | base line to fourth week
  MSK ultasound
craniovertebral angle | base line to fourth week
  angulus app to measure CVA

CONTACTS AND LOCATIONS:
Overall Officials: aisha razzaq, PHD, Principal Investigator — Riphah International University
Locations (1):
- Foundation University School of Health Sciences, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No